CLINICAL TRIAL: NCT01601171
Title: The Genetics of Neuroendocrine Reproductive Disorders and of the Cleft Lip and/or Palate
Brief Title: Genetics of Reproductive Disorders (Including Kallmann Syndrome) and Cleft Lip and/or Palate
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Nelly Pitteloud, Professor of Medicine, Chief of Service, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 345/11
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Kallmann Syndrome; Hypogonadotropic Hypogonadism; Hypothalamic Amenorrhea; Polycystic Ovarian Syndrome; Precocious Puberty; Cleft Lip and Palate; Cleft Palate; Cleft Lip
Keywords: GnRH deficiency; hypogonadism; anosmia; infertility; cleft lip; cleft palate; cryptorchidism; microphallus
MeSH Terms: conditions — Kallmann Syndrome; Hypogonadism; Polycystic Ovary Syndrome; Puberty, Precocious; Cleft Lip; Cleft Palate; Anosmia; Infertility; Cryptorchidism; Penis agenesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, serum/plasma, white blood cells, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with reproductive disorders with or without cleft lip/palate will be recruited for:
  * completion of medical questionnaire and review of medical records
  * family tree (including questions on reproductive disorders and cleft lip/palate)
  * specimen collection (DNA/RNA) from: serum/plasma/saliva/urine/buccal swab/hair follicles/sperm/skin biopsy
  * smell testing
  * hearing test
  * bone density
  * brain MRI
  * kidney, testicular/ovarian ultrasound
- Family members: Family members of Patients will be recruited for:
  * completion of medical questionnaire
  * specimen collection (DNA/RNA) from: serum/plasma/saliva/urine/buccal swab/hair follicles/sperm/skin biopsy
  * smell testing

SUMMARY:
The purpose of this study is to explore the genetic basis of reproductive disorders and cleft lip and/or palate.

DETAILED DESCRIPTION:
The World Health Organization estimates approximately 10% of couples experience some sort of infertility problem.

In humans, puberty is the process through which we develop reproductive capacity.

The timing of puberty varies greatly in the general population and is influenced by both genetic and environmental factors. In extreme cases of pubertal delay, puberty progresses only partially or not at all and results in the clinical picture of congenital hypogonadotropic hypogonadism (CHH), either accompanied by anosmia in 50% of cases (Kallmann syndrome [KS]) or by normal sense of smell (nCHH), with a male: female ratio of 4:1.

CHH is due to GnRH deficiency (incidence 1: 4,000-10,000) and result in the failure of sexual maturation and infertility. It is genetically heterogeneous, with multiple patterns of inheritance and several associated loci. In the clinical spectrum of GnRH deficiency, CHH may also be associated with a cleft lip/palate (CL/P) in 5 to 7% of cases. However, this prevalence increases up to 40% in CHH patients carrying a mutation in a CL/P gene, suggesting a genetic overlap between CHH and CL/P.

Disorders of puberty have provided insight into the biology of reproduction and genetic technologies have enabled us to deepen understanding in this field. The focus of this study is to better understand the genetic control of puberty and human reproduction as well as its link with CL/P.

Increasing understanding of the molecular basis (genes) of inherited reproductive disorders and CL/P may enable investigators to:

* improve diagnostic testing and treatments for these problems
* develop new diagnostic tests and therapies for patients
* enhance counseling for patients and families with reproductive disorders
* enhance counseling for patients and families with cleft lip/palate

ELIGIBILITY:
Inclusion Criteria:(any of the following conditions)

* hypogonadotropic hypogonadism
* Kallmann syndrome
* adult-onset hypogonadotropic hypogonadism
* hypothalamic amenorrhea
* polycystic ovarian syndrome
* primary gonadal failure
* precocious puberty
* cleft lip/palate
* family members of the above groups

Exclusion Criteria:

* acute illness/hospitalization
* pituitary tumors
* iron overload (hemochromatosis)
* infiltrative diseases (sarcoidosis)
* chronic alcohol abuse
* illicit drug use
* anabolic steroid abuse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be a convenience sample of those patients with reproductive disorders (and their family members), with or without cleft lip/palate, who are interested in participating in this genetic study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-03; Primary Completion 2025-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
rare sequence variant(s) in gene(s) | 1 year (ongoing if no variants are identified)
  The investigators aim to discover genes associated with reproductive disorders by identifying rare sequence variants (mutations) in patients

SECONDARY OUTCOMES:
functionality of identified rare sequence variants (mutations) | 1 year (following variant identification)
  The investigators will use a variety of scientific approaches to assess the functional impact of the identified rare sequence variants (mutations)
mode of inheritance | 1 year (following variant identification)
  The investigators will examine family pedigrees and study family members to determine the inheritance patterns (how the disorder is transmitted in the family)
genotype-phenotype correlation | 1 year (following variant identification)
  The investigators will study the phenotypic spectrum (how the disorder presents clinically) in patients with identified rare sequence variants (mutations)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Pitteloud, M.D., Principal Investigator — Centre Hositalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Miraoui H, Dwyer AA, Sykiotis GP, Plummer L, Chung W, Feng B, Beenken A, Clarke J, Pers TH, Dworzynski P, Keefe K, Niedziela M, Raivio T, Crowley WF Jr, Seminara SB, Quinton R, Hughes VA, Kumanov P, Young J, Yialamas MA, Hall JE, Van Vliet G, Chanoine JP, Rubenstein J, Mohammadi M, Tsai PS, Sidis Y, Lage K, Pitteloud N. Mutations in FGF17, IL17RD, DUSP6, SPRY4, and FLRT3 are identified in individuals with congenital hypogonadotropic hypogonadism. Am J Hum Genet. 2013 May 2;92(5):725-43. doi: 10.1016/j.ajhg.2013.04.008. PMID 23643382
- [Result] Villanueva C, Jacobson-Dickman E, Xu C, Manouvrier S, Dwyer AA, Sykiotis GP, Beenken A, Liu Y, Tommiska J, Hu Y, Tiosano D, Gerard M, Leger J, Drouin-Garraud V, Lefebvre H, Polak M, Carel JC, Phan-Hug F, Hauschild M, Plummer L, Rey JP, Raivio T, Bouloux P, Sidis Y, Mohammadi M, de Roux N, Pitteloud N. Congenital hypogonadotropic hypogonadism with split hand/foot malformation: a clinical entity with a high frequency of FGFR1 mutations. Genet Med. 2015 Aug;17(8):651-9. doi: 10.1038/gim.2014.166. Epub 2014 Nov 13. PMID 25394172
- See also: Web page for the Principal Investigator Nelly Pitteloud's research group — http://www.chuv.ch/edm/edm_home/edm-recherche/edm-research-groups/edm-researchgroup-pitteloud.htm